CLINICAL TRIAL: NCT01689116
Title: A Blinded Randomized Parallel Trial to Define the ECG Effects of Bardoxolone Methyl Using a Clinical and a Supratherapeutic Dose Compared to Placebo and Moxifloxacin (a Positive Control) in Healthy Men and Women: A Thorough ECG Trial.
Brief Title: Multiple-Dose Study of Effect of Bardoxolone Methyl on QT/QTC Interval Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-1006
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — bardoxolone methyl; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Bardoxolone Methyl 20mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl 20mg; Drug: Bardoxolone Methyl Placebo; Drug: Moxifloxacin Placebo
- Bardoxolone Methyl 80mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl 80mg; Drug: Moxifloxacin Placebo
- Bardoxolone Methyl Placebo (Placebo Comparator)
  Interventions: Drug: Bardoxolone Methyl Placebo; Drug: Moxifloxacin Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Bardoxolone Methyl Placebo; Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: Bardoxolone Methyl 20mg — Oral
  Arms: Bardoxolone Methyl 20mg
Drug: Bardoxolone Methyl 80mg — Oral
  Arms: Bardoxolone Methyl 80mg
Drug: Bardoxolone Methyl Placebo — Oral
  Arms: Bardoxolone Methyl 20mg; Bardoxolone Methyl Placebo; Moxifloxacin
Drug: Moxifloxacin 400mg — Oral
  Arms: Moxifloxacin
Drug: Moxifloxacin Placebo — Oral
  Arms: Bardoxolone Methyl 20mg; Bardoxolone Methyl 80mg; Bardoxolone Methyl Placebo

SUMMARY:
This is a single-center, multiple-dose, randomized, double-blind, double-dummy, placebo-controlled, active-comparator, parallel study in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet all of the following criteria to be included in the study:

1. Healthy male and female subjects between 18 to 50 years of age, inclusive. Healthy as determined by medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measurements performed at screening;
2. BMI greater than or equal to 18 kg/m2 but not to exceed 32 kg/m2;
3. Female subjects of childbearing potential must not be planning a pregnancy, pregnant, or lactating, and must have a negative serum pregnancy test result before enrollment into the study, and must be willing to use contraception as specified in section 12.8.3 or abstain from sexual activity for the duration of the study and for at least 3 weeks after discontinuation of study drug;
4. Male subjects and their partners of childbearing potential must use two methods of contraception, one of which must be a barrier method, for the duration of the study and for 30 days after completion;
5. Agree to abstain from alcohol consumption up to 3 days before dosing and throughout duration of the study (including the Study Day 13 visit);
6. Agree to abstain from strenuous exercise from 3 days before dosing and throughout duration of the study (including the Study Day 13 visit);
7. Able to effectively communicate with the investigator and other testing center personnel;
8. Able to participate, and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

All subjects with any of the following conditions or characteristics must be excluded from the study:

1. Currently participating in another study of an investigational drug (or a medical device) or have participated in another clinical study of an investigational drug (or a medical device) within 30 days of Study Day -1, 5 half-lives or twice the duration of biological effect of the previous investigational drug (whichever is longer);
2. Known hypersensitivity to any component in the formulation of the study drug, bardoxolone methyl;
3. Any medical or dental procedure, no matter how minor, that is planned or anticipated to occur during the conduct of the study;
4. History of drug or alcohol abuse or dependence within the last year;
5. History of smoking or tobacco use within the 6 months prior to Study Day -1;
6. Donation or receipt of blood or blood components within the 4 weeks prior to Study Day -1. The investigator should instruct subjects who participate in this study not to donate blood or blood components for 4 weeks after the completion of the study;
7. History of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or Torsades de Pointes, structural heart disease, or family history of long QT syndrome (suggested by sudden death due to cardiac causes at a young age of a close relative);
8. Evidence of any of the following cardiac conduction abnormalities based on the safety ECG at Screening:

   * Fridericia's correction for QT (QTcF) interval > 450 ms for males, > 470 ms for females;
   * PR interval < 110 ms or > 240 ms;
   * Intraventricular conduction delay with QRS duration >120 ms;
   * Resting heart rate < 40 bpm or > 90 bpm;
   * Pathological Q-waves (defined as Q-wave > 40 ms or depth > 0.4-0.5 mV);
   * Second- or third-degree atrioventricular block (AVB);
   * Electrocardiographic evidence of complete left bundle branch block (LBBB), right bundle branch block (RBBB), or incomplete left bundle branch block (LBBB);
   * Ventricular pre-excitation;
   * Atrial fibrillation, atrial flutter, or artificial cardiac pacemaker;
9. Screening ECG renders measurement of QT interval in lead II imprecise (for example: flat T waves, arrhythmias);
10. Subjects who have a screening supine blood pressure (BP) outside 90-145 mm Hg systolic or 45-95 mm Hg diastolic (measured following at least a 10-minute rest). Blood pressure may be re-tested twice in the supine position at intervals of 5 minutes. The pressure elevation is considered sustained if either the systolic or the diastolic pressure exceeds the stated limits after three assessments and the subject may not be randomized;
11. Use of any concomitant medications that are known to prolong QT/QTc interval within 30 days prior to Study Day -1;
12. Allergy to moxifloxacin or any fluoroquinolone antibiotic;
13. A positive test for drug(s) of abuse (alcohol, amphetamines, benzodiazepines, barbiturates, cocaine, opiates, or cannabinoids) at the screening or the Day -2 visit;
14. Any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the subject while involved in the study or could potentially influence the study outcome;
15. Positive test results for human immunodeficiency virus type 1 or 2 antibody at screening;
16. Any condition possibly affecting absorption, distribution, metabolism or excretion of drugs that may confound the analyses conducted in this study (for example: previous surgery on the gastrointestinal tract that includes removal of parts of stomach, bowel, liver, gall bladder, pancreas, venocaval shunts, or transjugular intrahepatic portosystemic shunts]);
17. Evidence or history of or concurrent clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dose administration), hematological, endocrine, immunological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease that in the judgment of the investigator could potentially either pose a health risk to the subject during the study or influence the study outcome;
18. Evidence of hepatic or biliary dysfunction including elevation of total bilirubin, direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), or alkaline phosphatase levels to greater than the upper limit of normal (ULN) at screening;
19. Abnormal hematological and biochemical parameters, including neutrophil count < 1500 cells/mm3, Hgb < 11 g/dL in females or < 12 g/dL in males, platelet count < 90,000 cells/mm3, creatinine ≥ 1.5 X ULN, albumin ≤ 3 g/dL, serum amylase or lipase ≥ 1.5X ULN at screening;
20. Positive test results for hepatitis B virus antibody, or hepatitis C virus antibody at screening;
21. Use of or need for any prescription or non-prescription systemic drug(s) including vitamins or herbal preparations other than drugs used for contraception, aspirin, acetaminophen, or other non-steroidal anti-inflammatory agents, within 10 days before Study Day -1 or during the study;
22. Use of aspirin, non-steroidal anti-inflammatory agents, or acetaminophen within 5 days prior to Study Day -1;
23. Consumption of alcohol- or caffeine-containing compounds within 24 hours before Day -2 visit;
24. Consumption of citrus juice within the 7 days before Day -2 visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Change in QT/QTc interval | Baseline, Day 6 and Day 13

SECONDARY OUTCOMES:
Maximum observed concentration | Day 1 and Day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Time to maximum observed concentration | Day 1 and Day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Area under the plasma concentration-time curve from time 0 to last observed concentration | Day 1 and Day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Area under curve for the dosing interval | Day 1 and Day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Accumulation index for maximum observed concentration | Day 1 and day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Accumulation index for area under the curve from time 0 to 24 hours | Day 1 and Day 6
  0 (immediately before dose administrations), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours following dose
Number of Adverse Events | Approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com
URL: https://vivli.org/